CLINICAL TRIAL: NCT02419339
Title: Prospective Multicenter Observational Study of Early Infancy Ureteral Reimplantation for Distal Ureteral Obstruction
Brief Title: Early Infancy Ureteral Reimplantation for Distal Ureteral Obstruction
Status: Terminated | Type: Observational
Why Stopped: Principal investigator is moving to a different institution.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0368-15-EP
Record Dates: First submitted 2015-04-08; First posted 2015-04-17 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Ureteral Obstruction; Urinary Diversion
MeSH Terms: conditions — Ureteral Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Extravesical ureteral reimplantation — Extravesical ureteral reimplantation with or without tapering

SUMMARY:
Prospective multicenter observational study of early infancy ureteral reimplantation for distal ureteral obstruction.

The study is an observation study since the investigators will not assign specific interventions to the subjects of the study.

The purpose of the study is to describe the surgical outcomes of early infancy ureteral reimplantation. Infants under 6 months of age with unilateral obstructed distal ureter, no other urologic pathologic and a normal contralateral kidney who have been recommended a ureteral reimplant by their pediatric urologist are eligible for the study. Patients that consent for the study will be prospectively followed for 1 year to record the outcomes of the surgery.

DETAILED DESCRIPTION:
Initial evaluation and determining if surgery is indicated:

Prenatal diagnosis: patient will get renal ultrasound at 2-7 days of birth and will be started on prophylaxis with amoxicillin or Keflex. At 6 weeks a VCUG, renal ultrasound and mag 3 will be done per local protocols.

Patients considered for reimplant will have:

1. SFU grade 3 and 4 hydroureteronephrosis
2. Normal contralateral kidney (VUR grade 1-3 ok) as defined above plus
3. Obstruction As defined by the BAPU (British Association of Paediatric Urologists consensus statement on the management of the primary obstructive megaureter)

If the patient meets criteria they will be consented for this observational study (before the surgery) and will have an extravesical ureteral reimplant in the next 0-2 months.

After the patient has been consented to participate in the study and before surgery, the investigators need to notify the main study site (Omaha) about the new patient and information will be recorded at the main site about the patient without patient identifiers. This is done so that they study can be analyze as an intention to treat.

Please note that this is an observational study: patients will have the same interventions and diagnostic tests regardless whether they chose or not to participate in the study. The investigator does not assign specific interventions to the subjects of the study. The protocol is only a suggested guideline to standardize details of the surgery and follow up of the patients among the different centers.

Postnatal diagnosis: patients with no history of prenatal hydronephrosis presenting with febrile UTI. If under 6 weeks of age they will be placed on prophylaxis with amoxicillin or Keflex. At 6 weeks a VCUG, renal ULTRASOUND and mag 3 will be done per local protocols. If presenting in between 6 weeks and 6 months of life they will undergo VCUG and Mag 3 after completing antibiotics course (7-10 days). Patients with febrile UTI not responding to antibiotics can be diverted with a percutaneous nephrostomy and once stable undergo testing.

Patients considered for reimplant will have:

1. SFU grade 3 and 4 hydroureteronephrosis
2. Normal contralateral kidney as defined above plus
3. Obstruction As defined by the BAPU If the patient fulfills criteria and the reimplant can be scheduled before age 7 months, they will be consented for the study.

After the patient has been consented to participate in the study and before surgery, the investigators need to notify the main study site (Omaha) about the new patient and information will be recorded at the main site about the patient without patient identifiers. This is done so that they study can be analyze as an intention to treat.

Patients initially not meeting criteria for surgery who had breakthrough UTI's Patients with unilateral megaureter but either no obstruction as defined above or no differential function loss can be considered for the study if they have Breakthrough UTI's while on prophylaxis and the surgery will be done at less than 7 months of age.

Follow up If patient does not meet criteria for surgery, follow up will be done as per local protocols with renal US +/- Mag 3 renal scans.

Follow up US can be done every 6-12 weeks. If US shows worsening patient can proceed with surgery or a Mag 3 can be done alternatively and any worsening >5% DFx on the mag 3 can could indicate surgery.

Below is a summary of patients eligible for surgery (all surgeries will have to be done under 7 months of age to enter into the study as well as inclusion and exclusion criteria must be followed):

1. Prenatally diagnosed unilateral distal obstruction that at 6 weeks have less than 40% DFx and SFU 3 or 4 hydronephrosis.
2. Patients who present postnatally with a febrile UTI and unilateral distal ureteral obstruction and on evaluation are found to have less than 40% DFx, and SFU 3 or 4 hydronephrosis.
3. Prenatally or postnatally diagnosed patients with distal obstruction who on initial evaluation did not meet criteria, but then subsequently had a Breakthrough febrile UTI's while on abx prophylaxis.
4. Prenatally or postnatally diagnosed patients with distal obstruction who on initial evaluation did not meet criteria, but on follow up US showed worsening hydronephrosis. Alternatively for these patients a Mag 3 can be repeated with surgery done for worsening parameters on the mag 3 (loss of more than 5% of function) .

Operative considerations Pfannenstiel incision. Fascial incision can be vertical or horizontal. Ureter dissected and divided at the bladder with 4-0 polydioxanone (suture ligation) if megaureter or as distal as possible/safe for ectopic ureter. Distal narrow or diseased looking segment excised.

Using 4 4-0 silk stay sutures, the borders or the detrusorrhaphy will be marked posterior laterally. A 3 cm detrusorrhaphy (minimum) down to mucosa will be done next.

Tapering (optional). Ureters more than 8-10 mm in diameter could be tapered. Based on some computer models research done by us, would recommend tapering just the distal ureter down to 4-5 mm in diameter over a stent left for 6 weeks. Ureter should not be tapered for more than a few centimeters in length to avoid devascularization. Alternatively, tapering can be left to the discretion of the surgeon.

The ureter will be anastomosed with running 5-0 or 6-0 polyglactin to the distal detrusorrhaphy making only a small mucosal opening.

A distal advancement suture will be placed to secure the UO distally in the bladder.

The detrusor will be then closed with interrupted 3-0 polyglactin stitches making sure no to obstruct the ureter proximal at the hiatus.

For non tapered reimplants, a stent will be sutured to the foley and removed in 5-7 days.

Drain at the discretion of the surgeon (preferably no drain) Foley will be left for 5-7 days in everyone. Overnight observation for all patients with extended hospital stay as needed for complications.

Follow up Antibiotic prophylaxis until first VCUG. (sulfamethoxazole/trimethoprim 3-4 mg/kg/day) 3 months: renal US, and VCUG. Mag 3 only for cases where the renal US showed no improvement (renal US stable or worse). Mag 3 can be done per the discretion of the surgeon too.

Continue antibiotic prophylaxis for girls and uncircumcised boys with VUR. May stop antibiotic prophylaxis for circumcised boy with VUR.

1 year: renal US, and VCUG (if previous VCUG showed VUR). Mag 3 only for cases where the renal US showed no improvement (renal US stable or worse). Mag 3 can be done per the discretion of the surgeon too.

Recurrent Febrile UTI's: will document any febrile UTI's defined at temp more than 38.5 with urine analysis with >10 white blood cells per high power field on microscopic exam and a positive urine culture more than 1 months after removal of foley or stent. Febrile UTI's within a month of the removal of foley or stent will be considered operative complications.

ELIGIBILITY:
Inclusion criteria:

* Children younger 6 months of age who have been recommended by their urologist to have a unilateral ureteral reimplant.
* Unilateral obstructive disease (as defined by the BAPU)
* Ipsilateral Single system
* Ipsilateral VUR is ok
* Contralateral reflux grades 1-3 ok as long as the reflux will be observed

Exclusion criteria

* Duplicated systems
* First Febrile UTI's and megaureter or ectopic ureter but no evidence of obstruction or loss of function
* Neurogenic bladder, valves
* Contralateral reflux grade 4-5

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants (under 6 months of age) undergoing an extravesical ureteral reimplant for primary obstructed megaureter or ectopic ureter.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Reoperation | 1 year
  Need for reoperation either for persistent documented obstruction or reflux with recurrent febrile UTI's

SECONDARY OUTCOMES:
Recurrent Febrile UTI's | 1 year
  Recurrent febrile urinary tract infections defined as fever more than 38.5, positive urine culture with more than 100,000 organism from a cath specimen and urine analysis with more than 10 leukocytes per high power field.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Villanueva, MD, Principal Investigator — University of Nebraska
Locations (1):
- Children's Hospital and Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] de Jong TP, Dik P, Klijn AJ, Uiterwaal CS, van Gool JD. Ectopic ureterocele: results of open surgical therapy in 40 patients. J Urol. 2000 Dec;164(6):2040-3; discussion 2043-4. PMID 11061921
- [Background] de Kort LM, Klijn AJ, Uiterwaal CS, de Jong TP. Ureteral reimplantation in infants and children: effect on bladder function. J Urol. 2002 Jan;167(1):285-7. doi: 10.1097/00005392-200201000-00084. PMID 11743341
- [Background] Gearhart JP. Primary obstructive ureter in neonates. Treatment by temporary uretero-cutaneostomy. Br J Urol. 1994 Jul;74(1):133-4. No abstract available. PMID 8044519
- [Background] Greenfield SP, Griswold JJ, Wan J. Ureteral reimplantation in infants. J Urol. 1993 Nov;150(5 Pt 1):1460-2. doi: 10.1016/s0022-5347(17)35809-3. PMID 8411425
- [Background] Kaefer M, Misseri R, Frank E, Rhee A, Lee SD. Refluxing ureteral reimplantation: a logical method for managing neonatal UVJ obstruction. J Pediatr Urol. 2014 Oct;10(5):824-30. doi: 10.1016/j.jpurol.2014.01.027. Epub 2014 Feb 28. PMID 24850437
- [Background] Kitchens DM, DeFoor W, Minevich E, Reddy P, Polsky E, McGregor A, Sheldon C. End cutaneous ureterostomy for the management of severe hydronephrosis. J Urol. 2007 Apr;177(4):1501-4. doi: 10.1016/j.juro.2006.11.076. PMID 17382764
- [Background] Kogan BA, Gohary MA. Cutaneous ureterostomy as a permanent external urinary diversion in children. J Urol. 1984 Oct;132(4):729-31. doi: 10.1016/s0022-5347(17)49844-2. PMID 6471219
- [Background] Lee SD, Akbal C, Kaefer M. Refluxing ureteral reimplant as temporary treatment of obstructive megaureter in neonate and infant. J Urol. 2005 Apr;173(4):1357-60; discussion 1360. doi: 10.1097/01.ju.0000152317.72166.df. PMID 15758801
- [Background] Liu C, Chin T, Wei C. Surgical treatment of vesicoureteral reflux in infants under 3 months of age. J Pediatr Surg. 1998 Nov;33(11):1716-9. doi: 10.1016/s0022-3468(98)90617-0. PMID 9856903
- [Background] MacGregor PS, Kay R, Straffon RA. Cutaneous ureterostomy in children--long-term followup. J Urol. 1985 Sep;134(3):518-20. doi: 10.1016/s0022-5347(17)47271-5. PMID 4032552
- [Background] Peters CA, Mandell J, Lebowitz RL, Colodny AH, Bauer SB, Hendren WH, Retik AB. Congenital obstructed megaureters in early infancy: diagnosis and treatment. J Urol. 1989 Aug;142(2 Pt 2):641-5; discussion 667-8. doi: 10.1016/s0022-5347(17)38842-0. PMID 2746792
- [Background] Sarduy GS, Crooks KK, Smith JP, Wise HA 2nd. Results in children managed by cutaneous ureterostomy. Urology. 1982 May;19(5):486-8. doi: 10.1016/0090-4295(82)90604-5. PMID 7080321
- [Background] Farrugia MK, Hitchcock R, Radford A, Burki T, Robb A, Murphy F; British Association of Paediatric Urologists. British Association of Paediatric Urologists consensus statement on the management of the primary obstructive megaureter. J Pediatr Urol. 2014 Feb;10(1):26-33. doi: 10.1016/j.jpurol.2013.09.018. Epub 2013 Oct 16. PMID 24206785